CLINICAL TRIAL: NCT06100744
Title: Open-label, Randomized, Assessor-blinded, Efficacy, Safety, Tolerability, and Pharmacokinetics Study of Subcutaneous Risankizumab With an Adalimumab Reference Arm in Children With Active Juvenile Psoriatic Arthritis
Brief Title: A Study to Assess Adverse Events, Change in Disease Activity, and How the Drug Moves Through the Body in Children With Juvenile Psoriatic Arthritis (jPsA) Receiving Subcutaneously Injected Risankizumab or Adalimumab
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M23-732; 2023-506026-36-00 (Other: EU CT)
Record Dates: First submitted 2023-10-20; First posted 2023-10-25 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Juvenile Psoriatic Arthritis
Keywords: Juvenile Psoriatic Arthritis; Psoriatic Arthritis; Risankizumab; ABBV-066; Adalimumab
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis, Psoriatic | interventions — Adalimumab; risankizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Risankizumab (Experimental): Participants will receive risankizumab for 24 weeks, in Period 1. Participants who respond to the study treatment received in Period 1, will continue to receive the same treatment in Period 2 for another 100 weeks. There will be a 140 day safety follow up after the treatment period.
  Interventions: Drug: Risankizumab
- Adalimumab (Experimental): Participants will receive adalimumab for 24 weeks, in Period 1. Participants who respond to the study treatment received in Period 1, will continue to receive the same treatment in Period 2 for another 100 weeks. There will be a 70 day safety follow up after the treatment period.
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — SC Injection
  Arms: Adalimumab
Drug: Risankizumab — Subcutaneous (SC) Injection
  Other Names: ABBV-066; Skyrizi
  Arms: Risankizumab

SUMMARY:
Psoriatic arthritis (PsA) is a type of arthritis that happens when the body's immune system attacks healthy cells and tissues causing joint pain, stiffness, and swelling. Symptoms can get worse and go away for periods of time. PsA that begins before a patient's 16th birthday is called juvenile PsA (jPsA).This study will evaluate how safe risankizumab is for the treatment of psoriatic arthritis and to assess change in disease symptoms.

Risankizumab is being studied for the treatment of jPsA and adalimumab is approved for the treatment of jPsA. Participants are placed in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 4 chance that participants will be assigned to receive adalimumab. Approximately 40 juvenile participants with jPsA will be enrolled at approximately 30 sites worldwide.

Participants will receive risankizumab and adalimumab as subcutaneous (SC) injections based on body weight. At the start of Period 1, participants are randomized to receive risankizumab or adalimumab for 24 weeks. Participants who respond to the study treatment received in Period 1, will continue to receive the same treatment in Period 2 for another 100 weeks. Those with worsening jPsA symptoms in Period 2 will be withdrawn from the study. Participants who receive adalimumab are followed for safety for 70 days after the last study treatment. Participants who receive risankizumab are followed for 140 days after the last study treatment.

There may be higher treatment burden for participants in this trial compared to their standard of care (due to study procedures). Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of juvenile psoriatic arthritis (jPsA) according to International League of Associations for Rheumatology criteria for at least 3 months prior to screening.
* Active Disease in >= 3 joints at screening and at Baseline (swelling not due to deformity, or limitation of motion with pain, tenderness, or both) are eligible for inclusion in the study.
* Have had an inadequate response (lack of efficacy after minimum 2-month duration of therapy at maximally tolerated dose), or intolerance to previous or current treatment with at least 1 of the following conventional synthetic disease-modifying antirheumatic drug (csDMARDs): methotrexate (MTX), sulfasalazine, leflunomide, or hydroxychloroquine.

Exclusion Criteria:

* Have any other autoimmune disease, rheumatic disease (including systemic Juvenile idiopathic arthritis [JIA], rheumatoid factor-positive or rheumatoid factor-negative polyarticular JIA, extended oligoarticular JIA, persistent oligoarticular JIA, enthesitis-related arthritis, and undifferentiated JIA), or overlap syndrome.
* Prior inadequate response to treatments in the anti-TNF or IL-23 inhibitor classes.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants who Achieve >= 30% Improvement in Juvenile Idiopathic Arthritis American College of Rheumatology Response Criteria (JIA-ACR 30) | Up to 24 Weeks
  The JIA-ACR 30 response is defined as a >= 30% improvement of at least 3 or more of the 6 juvenile idiopathic arthritis core response variables (JIA-CRVs) without >30% worsening in more than 1 of the remaining JIA-CRVs compared with Baseline. The 6 JIA-CRVs are: physician global assessment of disease activity (PhGA), global assessment of overall well being, no of joints with active arthritis, no of joints with limitation of motion high sensitivity C-reactive protein (hsCRP), and functional ability assessed by Childhood Health Assessment Questionnaire Disability Index (CHAQ-DI).
Number of Participants with Adverse Events (AEs) | Up to Week 144
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants who Achieve >= 50% Improvement in Juvenile Idiopathic Arthritis American College of Rheumatology Response Criteria (JIA-ACR 50) | Up to 24 Weeks
  The JIA-ACR 50 response is defined as a >= 50% improvement of at least 3 or more of the 6 JIA-CRVs without >50% worsening in more than 1 of the remaining JIA-CRVs compared with Baseline. The 6 JIA-CRVs are: PhGA, parent/patient global assessment of overall well being, no of joints with active arthritis, no of joints with limitation of motion hsCRP, and functional ability assessed using the disability index of the CHAQ-DI.
Percentage of Participants who Achieve >= 70% Improvement in Juvenile Idiopathic Arthritis American College of Rheumatology Response Criteria (JIA-ACR 70) | Up to 24 Weeks
  The JIA-ACR 70 response is defined as a >= 70% improvement of at least 3 or more of the 6 JIA-CRVs without >70% worsening in more than 1 of the remaining JIA-CRVs compared with Baseline. The 6 JIA-CRVs are: PhGA, parent/patient global assessment of overall well being, no of joints with active arthritis, no of joints with limitation of motion hsCRP, and functional ability assessed using the disability index of the CHAQ-DI.
Percentage of Participants who Achieve >= 90% Improvement in Juvenile Idiopathic Arthritis American College of Rheumatology Response Criteria (JIA-ACR 90) | Up to 24 Weeks
  The JIA-ACR 90 response is defined as a >= 90% improvement of at least 3 or more of the 6 JIA-CRVs without >90% worsening in more than 1 of the remaining JIA-CRVs compared with Baseline. The 6 JIA-CRVs are: PhGA, parent/patient global assessment of overall well being, no of joints with active arthritis, no of joints with limitation of motion hsCRP, and functional ability assessed using the disability index of the CHAQ-DI.
Change from Baseline in Juvenile Arthritis Disease Activity Score (JADAS)-10 | Up to Week 24
  JADAS is a composite score of physician global assessment of disease activity, parent/patient global assessment of overall well-being, number of joints with active arthritis (swelling not due to deformity, or limitation of motion with pain, tenderness or both), and high sensitivity C-reactive protein (hsCRP). JADAS-10 is based on the count of any involved joint, up to a maximum of ten joints.
Change from Baseline in JADAS-27 | Up to Week 24
  JADAS is a composite score of physician global assessment of disease activity, parent/patient global assessment of overall well-being, number of joints with active arthritis (swelling not due to deformity, or limitation of motion with pain, tenderness or both), and hsCRP. JADAS-27 includes a count of the following joints: cervical spine, elbows, wrists, metacarpophalangeal joints (from first to third), and proximal interphalangeal joints, hips, knees, and ankles.
Percentage of Participants with Achievement of Minimal Disease Activity (MDA) | Week 24
  MDA is defined as JADAS-10 of <= 6. JADAS-10 is based on the count of any involved joint, up to a maximum of ten joints.
Percentage of Participants with Inactive Disease | Week 24
  Inactive disease is defined as JADAS-10 of <= 2.7. JADAS-10 is based on the count of any involved joint, up to a maximum of ten joints.
Change from Baseline in Clinical Juvenile Arthritis Disease Activity Score (cJADAS)-10 | Up to Week 24
  cJADAS is a composite score of physician global assessment of disease activity, parent/patient global assessment of overall well-being, and number of joints with active arthritis (swelling not due to deformity, or limitation of motion with pain, tenderness or both). JADAS-10 is based on the count of any involved joint, up to a maximum of ten joints.
Change from Baseline in cJADAS-27 | Up to Week 24
  cJADAS is a composite score of physician global assessment of disease activity, parent/patient global assessment of overall well-being, and number of joints with active arthritis (swelling not due to deformity, or limitation of motion with pain, tenderness or both). JADAS-27 includes a count of the following joints: cervical spine, elbows, wrists, metacarpophalangeal joints (from first to third), and proximal interphalangeal joints, hips, knees, and ankles.
Change from Baseline in the Pain-Visual Analogue Scale (VAS) | Week 24
  Participants assessed their pain using a Patient's Global Assessment Pain visual analogue scale (VAS). The range is 0 to 100 with no pain being indicated by 0 and severe pain by 100.
Percentage of Participants with Psoriasis (PsO) who Achieve Psoriasis Area Severity Index (PASI) 75 in Participants with at least 3% Body Surface Area (BSA) at Baseline | Up to Week 24
  The PASI is a measure of psoriasis severity. Four anatomic sites - head, upper extremities, trunk, and lower extremities - are assessed for erythema, induration and desquamation using a 5-point scale, with a lower score indicating more mild disease.
Percentage of Participants with PsO who Achieve PASI 90 in Participants with at least 3% BSA at Baseline | Up to Week 24
  The PASI is a measure of psoriasis severity. Four anatomic sites - head, upper extremities, trunk, and lower extremities - are assessed for erythema, induration and desquamation using a 5-point scale, with a lower score indicating more mild disease.
Percentage of Participants with PsO who Achieve Static Physician Global Assessment of Disease Activity (sPGA) of PsO of 'Clear' (0) or Almost Clear (1) in Participants with at least 3% BSA at Baseline | Up to Week 24
  The sPGA is a 5-point score ranging from 0 to 4, based on the physician's assessment of the average thickness, erythema, and scaling of all psoriatic lesions, with a lower score indicating less body coverage.
Percentage of Participants with PsO who Achieve change from Baseline in Children's Dermatology Life Quality Index (CDLQI) in Participants with at least 3% BSA at Baseline | Up to Week 24
  The CDLQI is a 10-item questionnaire used to assess the impact of dermatologic disease symptoms and treatment on quality-of-life (QOL), with a higher score indicating greater impairment of QOL. The CDLQI has been validated for use in participants 4 to 16 years old.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (31):
- United States (9):
  - Arkansas Children's Hospital /ID# 258776, Little Rock, Arkansas
  - Childrens National Medical Center /ID# 259284, Washington D.C., District of Columbia
  - Joe Dimaggio Children's Hospital Hollywood /ID# 260634, Hollywood, Florida
  - Indiana University Health Riley Hospital for Children /ID# 259067, Indianapolis, Indiana
  - M Health Fairview University of Minnesota Medical Center - West Bank /ID# 260111, Minneapolis, Minnesota
  - Boston Childrens Health Physicians /ID# 258061, Valhalla, New York
  - University of North Carolina - Children's Hospital /ID# 259286, Chapel Hill, North Carolina
  - MetroHealth Medical Center /ID# 262377, Cleveland, Ohio
  - Child Neurology Consultants of Austin /ID# 260562, Austin, Texas
- Monash Health - Monash Medical Centre /ID# 260255, Clayton, Victoria, Australia
- Canada (3):
  - Alberta Children's Hospital /ID# 257880, Calgary, Alberta
  - British Columbia Children and Women's Hospital and Health Centre /ID# 257884, Vancouver, British Columbia
  - Hospital for Sick Children /ID# 257879, Toronto, Ontario
- France (2):
  - CHU Bordeaux - Hopital Pellegrin /ID# 258729, Bordeaux, Nouvelle-Aquitaine
  - AP-HP - Hopital Bicetre /ID# 258728, Le Kremlin-Bicêtre, Paris
- Germany (3):
  - Asklepios Klinik Sankt Augustin /ID# 259106, Sankt Augustin, North Rhine-Westphalia
  - Helios Klinikum Berlin - Buch /ID# 268803, Berlin
  - Hamburger Zentrum fuer Kinder- und Jugendrheumatologie /ID# 259104, Hamburg
- Italy (3):
  - Azienda Ospedaliero Universitaria Meyer /ID# 258587, Florence, Firenze
  - ASST Centro Specialistico Ortopedico Traumatologico Gaetano Pini-CTO /ID# 276753, Milan, Milano
  - Ospedale Pediatrico Bambino Gesù /ID# 258869, Rome, Roma
- Poland (5):
  - Malopolskie Badania Kliniczne /ID# 258777, Krakow, Lesser Poland Voivodeship
  - Uniwersytecki Szpital Dzieciecy w Lublinie /ID# 258781, Lublin, Lublin Voivodeship
  - Narodowy Instytut Geriatrii, Reumatologii I Rehabilitacji /ID# 277050, Warsaw, Masovian Voivodeship
  - Centrum Zdrowia Dziecka i Rodziny im Jana Pawla II w Sosnowcu /ID# 277058, Sosnowiec, Silesian Voivodeship
  - SPZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi /ID# 258785, Lodz, Łódź Voivodeship
- Spain (2):
  - Hospital Sant Joan de Deu /ID# 257568, Esplugues de Llobregat, Barcelona
  - Hospital Universitario y Politecnico La Fe /ID# 257567, Valencia
- United Kingdom (3):
  - Sheffield Children's Hospital NHS Foundation Trust /ID# 258848, Sheffield, England
  - University Hospitals Bristol and Weston NHS Foundation Trust /ID# 258847, Bristol
  - Alder Hey Children's NHS Foundation Trust /ID# 262770, Liverpool

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-732